CLINICAL TRIAL: NCT01797848
Title: A Phase 3 Randomized, Double Blind, Multi-National Evaluation of Daclatasvir in Combination With Peg Interferon Alfa-2a and Ribavirin in Treatment-Naive Subjects With Chronic Hepatitis C Genotypes 1 and 4
Brief Title: Efficacy and Safety Evaluation of a Treatment Consisting of Peg Interferon Alfa + Ribavirin + Daclatasvir in HCV Genotype 1 and 4 Treatment naïve Patients
Acronym: COMMAND-Asia
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AI444-047
Record Dates: First submitted 2013-02-21; First posted 2013-02-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon alfa-2a; Ribavirin; daclatasvir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- pegIFNα 2a + Ribavirin + Placebo (Experimental): pegIFNα 2a 180 µg, Solution for injection, Subcutaneous, Once weekly, 48 weeks
  Ribavirin 200 mg Tablets, by mouth, 400-600mg AM, 600 mg PM, 48 weeks
  Placebo 0 mg Tablets, by mouth, Once daily, 24 weeks
  Interventions: Drug: Peginterferon alfa 2a; Drug: Ribavirin; Drug: Placebo matching Daclatasvir
- pegIFNα 2a + Ribavirin + Daclatasvir (Experimental): pegIFNα 2a 180 µg, Solution for injection, Subcutaneous, Once weekly, 24 or 48 weeks depending on response
  Ribavirin 1000-1200 mg Tablets, by mouth, 400-600mg AM, 600 mg PM, 24 or 48 weeks depending on response
  Daclatasvir 60 mg Tablets, by mouth, Once daily, 24 weeks
  Interventions: Drug: Peginterferon alfa 2a; Drug: Ribavirin; Drug: Daclatasvir

INTERVENTIONS:
Drug: Peginterferon alfa 2a
  Other Names: Pegasys®
Drug: Ribavirin
  Other Names: Copegus® (Taiwan, Korea and Singapore); Wei Lining (China)
Drug: Placebo matching Daclatasvir
  Arms: pegIFNα 2a + Ribavirin + Placebo
Drug: Daclatasvir
  Other Names: BMS-790052-05
  Arms: pegIFNα 2a + Ribavirin + Daclatasvir

SUMMARY:
The purpose of this study is to determine whether 24 week treatment with the Daclatasvir (DCV) in combination with Pegylated-interferon alfa 2a (pegIFNα-2a) and Ribavirin (RBV) is safe and demonstrates rate of Sustained Virologic Response at follow up week 24 (SVR24) (defined as undetectable HCV RNA at post-treatment Week 24) that are non-inferior to 48 weeks of the dual combination therapy of pegIFNα-2a/RBV in a majority of study subjects

ELIGIBILITY:
Inclusion Criteria:

* Patients chronically infected with Hepatitis C virus (HCV) GT 1 or 4
* HCV RNA viral load ≥ 10,000 IU/mL
* Naïve to prior treatment with any interferon formulation, Ribavirin (RBV) or HCV direct antiviral agent
* Patients with compensated cirrhosis are permitted

Exclusion Criteria:

* Infected with HCV other than GT 1 or 4
* Evidence of decompensated liver disease
* Documented or suspected Hepatocellular carcinoma (HCC) as evidenced by previously obtained imaging studies or liver biopsy
* Evidence of a medical condition contributing to chronic liver disease other than HCV
* History of chronic Hepatitis B virus (HBV) or Human immunodeficiency virus (HIV)
* Current or know history of cancer (except in situ carcinoma of cervix or adequately treated basal or squamous cell carcinoma of the skin) within 5 years prior to enrollment
* Laboratory values:

  1. Hemoglobin < 12 g/dL (females) or < 13 g/dL (males)
  2. Platelets < 90 x 1000000000 cells/L
  3. Absolute neutrophil count (ANC) < 1.5 × 1000000000 cells/L
  4. Total bilirubin ≥ 34 µmol/L (unless due to Gilbert's disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of Genotype 1 subjects with SVR24, defined as HCV RNA < Limit of quantification (LOQ) at follow-up Week 24 for each cohort | Week 24 post treatment follow up

SECONDARY OUTCOMES:
Proportion of Genotype (GT) 4 subjects with SVR24 | Week 24 post treatment follow up visit
Proportion of GT 1 & 4 subjects who achieve HCV RNA < LOQ or undetectable | Week 24 post treatment follow up visit and Week 48 post treatment follow up visit for subjects who achieve Virologic response [VR] (4&12)
Frequency of Serious Adverse Events (SAEs)/discontinuations due to Adverse Events (AEs) | Up to 48 weeks plus 30 days
Discontinuations due to Adverse Events (AEs) | Up to 48 weeks plus 7 days
Proportion of subjects with Sustained Virologic Response at follow up week 12 (SVR12) or SVR24 by rs12979860 Single nucleotide polymorphism (SNP) in the IL28B gene | Up to 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx